CLINICAL TRIAL: NCT02032706
Title: Validation of Safety and Efficacy for Night Shift Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Brain Monitoring, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201301
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2014-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; position therapy; snoring; positional
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positional feedback (Experimental): Deliver therapy when the supine position is detected
  Interventions: Device: Deliver therapy when the supine position is detected

INTERVENTIONS:
Device: Deliver therapy when the supine position is detected — Application of vibrotactile feedback to the neck when the supine position is detected
  Other Names: Night Shift

SUMMARY:
The purpose of this study is to assess the accuracy of Night Shift in the detection of supine sleep and efficacy of vibro-tactile feedback in restricting supine sleep.

DETAILED DESCRIPTION:
The protocol is designed to first evaluate the accuracy of supine vs. non-supine detection in 15 subjects (hereafter referred to as study 1). In study 2, patients who had completed a baseline polysomnography (PSG) with a minimum of four hours of sleep time were to wear the Night Shift for two nights without feedback to confirm their willingness to continue with the study, followed by 28 nights of vibro-tactile position therapy. A follow-up PSG was to be conducted as soon as possible to the completion of the 28-nights of treatment. During enrollment subjects were to complete pre-treatment questionnaires designed to measure daytime sleepiness, insomnia severity, depression, anxiety, and quality of life. The same instruments were completed post-treatment on the morning after the 28th night of treatment. Subjects completed daily logs to confirm device utilization and identify potential non-device related factors that could influence study completion.

ELIGIBILITY:
The inclusion criteria are:

* be between the age of 18 and 75 years,
* have been diagnosed with Obstructive Sleep Apnea (OSA) during polysomnography at a designated sleep center within 4 months of their enrollment,
* have not received treatment with any OSA therapy for more than 3 days within the past month,
* have an overall Apnea-Hypopnea Index (AHI) > 10 and hypopneas requiring >3% oxygen desaturation,
* having a non-supine Apnea-Hypopnea Index (AHI) < 15 if Continuous Positive Airway Pressure has not been attempted,
* have a overall AHI divided by the non-supine AHI > 1.5,
* had an Epworth Sleepiness Score of 5 or more at the time of diagnosis and at the start of therapy,
* Change in weight of no more than 5 pounds since the diagnostic PSG
* access to a computer and the Internet
* sleep is sometime between 8 P.M. to 9 A.M. Monday through Friday in the same bed

Exclusion Criteria:

* Neck, back or should pain which would impact ability to sleep laterally each night
* Body mass index > 35
* suffering from neurological disorders which result in ticks or tremors
* diagnosed with congestive heart failure or chronic obstructive pulmonary disease
* suffered from a stroke within the previous 12 months
* taking or planning to take narcotic medications
* unfamiliar with use of internet browsers
* travel (i.e., foreign or cruise ship) which would limit internet or mail access
* planned medical procedures (e.g., surgery) which would limit device use during the scheduled 30-day study period or introduce the need for narcotic pain medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Levendowski, MBA, Principal Investigator — Advanced Brain Monitoring, Inc.
Locations (1):
- Complete Sleep Solutions, Murrieta, California, United States

REFERENCES:
- [Background] Levendowski DJ, Seagraves S, Popovic D, Westbrook PR. Assessment of a neck-based treatment and monitoring device for positional obstructive sleep apnea. J Clin Sleep Med. 2014 Aug 15;10(8):863-71. doi: 10.5664/jcsm.3956. PMID 25126032
- [Background] Levendowski DJ, Veljkovic B, Seagraves S, Westbrook PR. Capability of a neck worn device to measure sleep/wake, airway position, and differentiate benign snoring from obstructive sleep apnea. J Clin Monit Comput. 2015 Feb;29(1):53-64. doi: 10.1007/s10877-014-9569-3. Epub 2014 Mar 6. PMID 24599632
- See also: Related Info — http://advancedbrainmonitoring.com/night-shift/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positional Feedback
Started | 36
Completed | 30
Not Completed | 6
Not completed — Did not qualify | 5
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: 36 subjects were studied at baseline, 5 were dropped due to not meeting the required continuation criteria, 1 was dropped due to not following the protocol requirements. Follow-up PSG studies were conducted and data are available from the 30 participants who completed the study.
Arm/Group | Positional Feedback
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Completed the Study at 4 Weeks Without Adverse Events
Description: Assess the potential for adverse events by evaluating whether more than 20% of participants chose to terminate the study prior to completing 4 weeks of therapy.
Time Frame: Four weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Positional Feedback
Number analyzed (Participants) | 30
Percentage of participants | 100

2. Primary Outcome: Evaluate Efficacy Based on a Change in Obstructive Sleep Apnea (OSA) Severity as a Result of Therapy
Description: Determine the percentage of participants that exhibited at least a 50% reduction in OSA severity measured by AHI after 4 weeks of therapy.
Time Frame: 30-days
Measure: Number; unit: percentage of participants
Arm/Group | Positional Feedback
Number analyzed (Participants) | 30
percentage of participants | 83

3. Secondary Outcome: Confirmation That Night Shift Accurately Detects Supine Position
Description: Compute the percentage of participants at baseline and at followup in which the Night Shift's measurement of the supine position was within+/- 5% of the percent time supine by video recordings plus chest sensor (gold standard).
Time Frame: baseline and 4-weeks later at follow up
Population: 35 subjects completed the baseline polysomnography (PSG) while wearing the device. One subject's PSG study was conducted prior to enrollment but qualified as a baseline. 30 subjects completed a follow-up PSG.
Measure: Number; unit: percentage of participants
Arm/Group | Positional Feedback
Number analyzed (Participants) | 35
percentage of participants
  Baseline accuracy n=35 | 91
  Followup accuracy n=30 | 93

4. Secondary Outcome: Evaluate Whether Night Shift Disrupts Sleep Such That Users Are Non-compliant
Description: Measure the percentage of nights across the 4 weeks of therapy the Night Shift was worn for a minimum of 5.5 hours/night or the length of time in bed by each participant.
Time Frame: four weeks
Measure: Median (Full Range); unit: Percent of nights
Arm/Group | Positional Feedback
Number analyzed (Participants) | 30
Percent of nights | 96 [71 to 100]

5. Secondary Outcome: Evaluate Whether Patients Adapt and Sleep Through the Position Therapy Feedback
Description: Evaluate the percent time supine across four weeks of use and confirm that participants average less than 15% time supine across the four weeks of home use
Time Frame: four weeks
Measure: Number; unit: % participants averaged < 15% supine
Arm/Group | Positional Feedback
Number analyzed (Participants) | 30
% participants averaged < 15% supine | 97

6. Secondary Outcome: Evaluate Efficacy by Confirming Position Therapy Reduces Daytime Somnolence in Patients With Positional OSA
Description: The percentage of compliant participants who show an improved Epworth Sleepiness Score of >= 2 after 4 weeks of therapy when compared to the baseline score. Epworth scores range from 0 (no daytime somnolence) to 21 being extreme somnolence. A difference of 2 or more indicates some positive benefit from therapy.
Time Frame: baseline and followup
Measure: Number; unit: percentage of participants
Arm/Group | Positional Feedback
Number analyzed (Participants) | 30
percentage of participants | 50

7. Secondary Outcome: Evaluate Impact of Positional Therapy on Quality of Life Scores
Description: Compare the Functional Outcomes of Sleep (FOSQ) scores obtained at baseline and compare to results after 4 weeks of therapy to determine the percentage of compliant participants who demonstrate >2 point improvement. The FOSQ includes thirty questions with numerically scaled responses which are totaled with an overall score of 1 identifying the most impaired and 120 identifying the least impaired.
Time Frame: four weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Positional Feedback
Number analyzed (Participants) | 30
Percentage of participants | 57

8. Secondary Outcome: Assess the Accuracy of Night Shift's Detection of Sleep vs. Wake
Description: Compare the epochs staged wake and sleep by the reference standard (polysomnography) to the epochs staged wake and sleep by Night Shift to determine the sleep (sensitivity) and wake (specificity) classification accuracy.
Time Frame: baseline and follow-up
Measure: Mean (Standard Deviation); unit: percentage of epochs
Arm/Group | Positional Feedback
Number analyzed (Participants) | 35
percentage of epochs
  Sensitivity sleep baseline | 88.7 (8.9)
  Sensitivity sleep followup | 91.3 (8.0)
  Specificity wake baseline | 55.0 (17.7)
  Specificity wake followup | 61.2 (16.5)

9. Secondary Outcome: Assess the Accuracy of Night Shift's Measurement of Total Sleep Time
Description: Compared the Total Sleep Time (TST) from polysomnography to the Night Shift TST to tally the number of records with differences outside the range (151 to -129) defined by the predicate device.
Time Frame: one night
Population: Comparisons included 35 studies at baseline and 30 follow-up studies
Measure: Number; unit: % of studies
Arm/Group | Positional Feedback
Number analyzed (Participants) | 35
% of studies | 98

10. Secondary Outcome: Assess the Accuracy of Night Shift Measurement of Sleep Efficiency
Description: Compare Sleep Efficiency (SE) obtained from PSG and compared to the Night Shift SE to determine if outliers are within the range (19.1 to -17.2%) defined by the predicate device
Time Frame: one night
Population: Studies included 35 baseline comparisons and 30 comparisons at follow-up
Measure: Number; unit: % studies
Arm/Group | Positional Feedback
Number analyzed (Participants) | 35
% studies | 92

ADVERSE EVENTS:
Time Frame: Throughout the study duration i.e., four weeks of use
Arm/Group | Positional Feedback
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No